CLINICAL TRIAL: NCT04367558
Title: Possible Efficacy of Minimal Surgical Treatment for Obstructive Sleep Apnea (OSA)
Brief Title: Minimal Surgical Treatment for Obstructive Sleep Apnea (OSA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0010-20-HYMC
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Sleep Apnea Syndromes, Obstructive
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Patient suffering from OSA, and found to suffer from obstruction of one or more of the following areas - Lower turbines, Soft Palate, Tonsils, Base-of-tongue.
  Interventions: Procedure: Minimally invasive, in-office, RF reduction of the affected area

INTERVENTIONS:
Procedure: Minimally invasive, in-office, RF reduction of the affected area — Usage of RF needle to treat one or more of the affected areas

SUMMARY:
Obstructive Sleep apnea carries a variety of complications and implications. While the disease could be treated using continuous positive airway pressure (CPAP) and lifestyle changes, many patients find it difficult to adjust to the mask, and turn to surgical options. The conventional surgical options to date ranges from radical (UPPP) to individualized, with or without Drug-induced sleep endoscopy (DISE). Previous studies showed that dise directed surgery can be useful for specific conditions. No trials were found to test in-office encompassing minimal invasive surgical treatment (RF palatoplasty , RF tonsillotomy, RF turbinectomy, and RF base-of-tongue reduction) as a viable alternative..

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from OSA, defined as AHI > 5

Exclusion Criteria:

* Patients who can use CPAP.
* Patients suffering from confounding factors with higher risk (Coagulation problems, Heart conditions, chronic obstructive pulmonary disease (COPD), or other dangerous conditions as decided by the surgeon)
* Patients suffering from other problems aggravating the OSA (Respiratory, Neurologic conditions)

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
More than 50% improvement in Apnea-Hypopnea index (AHI) | 6 months following the procedure
  Measuring the AHI score using sleep laboratory
More than 50% improvement in Apnea-Hypopnea index (AHI) | 12 months following the procedure
  Measuring the AHI score using sleep laboratory
Reduction of AHI to below 20 | 6 months following the procedure
  Measuring the AHI score using sleep laboratory
Reduction of AHI to below 20 | 12 months following the procedure
  Measuring the AHI score using sleep laboratory

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe MC,, Hadera, Israel

IPD SHARING:
Plan to Share IPD: Undecided